CLINICAL TRIAL: NCT05498623
Title: MR Fingerprinting of the Prostate - Towards Improved Patient Care with High Speed Quantitative Imaging
Brief Title: MR Fingerprinting for Diagnostic of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 218665
Record Dates: First submitted 2022-07-05; First posted 2022-08-12 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Magnetic Resonance Imaging
Keywords: MR Fingerprinting; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The diagnostic pathway for suspected prostate cancer relies greatly on radiological imaging. Establishment of magnetic resonance fingerprinting (MRF) has the potential to significantly improve patient experience and outcomes. MRF is a novel and innovative approach to a long-standing challenge of recording and reconstructing MR image

The aim is to conduct a clinical pilot study in which patients will be scanned using the newly refined MRF sequence in addition to the conventional scanning protocols.

DETAILED DESCRIPTION:
The patient is at the center of all medical interventions and innovations. For those with prostate cancer, the pathway for new patients has scope for improvement. MRI is an important and necessary part of that pathway, but scanning capacity is often stretched, and there is need for effective and efficient scan techniques. Beyond mere detection of lesions, the modality has potential to differentiate and categorize the clinical significance of prostate cancer. By virtue of quantitative imaging, the determination of biomarkers could lead to a non-invasive method of prostate cancer diagnosis. The Prostate Imaging Reporting and Data System (PIRADS) scoring is a standardized system of acquiring and categorizing multi-parametric-MR images (mp-MRI) of the prostate. The PIRADS system works to grade to clinical significance of prostate cancer, however this relies on qualitative information.

Patients referred for a typical MRI of the prostate will in addition receive the MR Fingerprinting scan, which will add about 8 minutes to their time on the scanner. The direct comparison of the fingerprint maps and multi-parametric images can then be made. Conclusions will be drawn with focus to potential improvement of the PIRADS protocol.

The main aim of the project is therefor to implement, validate, and optimize sequences for MR Fingerprinting of the prostate.

ELIGIBILITY:
Inclusion Criteria:

- Men referred to an MR examination for prostate cancer diagnostic

Exclusion Criteria:

- None

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited among students and employees at NTNU/St. Olavs Hospital. The possibility to participate will be announced on internal WEB-pages and on bulletin boards at Øya Campus.
  Patients referred to mp-MRI due to suspicion of prostate cancer will receive information about the study and the informed consent form together with the letter they receive from Clinic of Radiology with their appointment for the MRI examination.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
MRF compared to T1, T2 and proton density generated to the PIRADS scoring | an average of 30 minutes
  MR Fingerprinting has proven to reduce scan time by acquiring property maps simultaneously. MRF uses pseudorandom, rapidly switching pulses to elicit a unique signal evolution - hence the term fingerprint. This "fingerprint" signal is matched to a predefined dictionary of all possible signal evolutions and so multiple measurements are acquired simultaneously. Since the values such as T1, T2 and proton density are matched and not interpolated, the method is far more quantitative than conventional MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Ma D, Gulani V, Seiberlich N, Liu K, Sunshine JL, Duerk JL, Griswold MA. Magnetic resonance fingerprinting. Nature. 2013 Mar 14;495(7440):187-92. doi: 10.1038/nature11971. PMID 23486058
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566